CLINICAL TRIAL: NCT01807299
Title: The Effect of Physical Training and the Omega 3 Consumption on Attention Deficit
Brief Title: The Effect of Physical Training and the Omega 3 Consumption on Attention Deficit Hyperactivity Disorder in Children
Acronym: AOE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Fernandes Galduroz MD, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADHD_Omega_Exercise
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Physical Training; ADHD-Attention deficit hyperactivity disorder; Omega 3
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Docosahexaenoic Acids; Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Physical Training (Experimental): The training group will make physical exercise for three months (three times a week).
  Interventions: Dietary Supplement: Omega 3
- Sedentary (Other): The sedentary group will be oriented not to make any type of physical training for three months.
  Interventions: Dietary Supplement: Omega 3
- Placebo (Placebo Comparator): The omega 3 group will receive 2g per day of mineral oil during 90 days treatment
  Interventions: Other: Physical Training
- Omega 3 (Experimental): The omega 3 group will receive 2g per day of fish oil during 90 days treatment
  Interventions: Other: Physical Training

INTERVENTIONS:
Dietary Supplement: Omega 3 — Capsules of omega 3, 1000mg / capsules. Administered 3 times a day.
  Arms: Physical Training; Sedentary
Other: Physical Training
  Arms: Omega 3; Placebo

SUMMARY:
The attention deficit hyperactivity disorder (ADHD) usually occurs in preschool and may cause disabilities through whole life.

DETAILED DESCRIPTION:
The attention deficit hyperactivity disorder (ADHD) usually occurs in preschool and may cause disabilities through whole life. The treatment of this disease is expensive and difficult. Moreover, physical exercise and omegas consumption may improve the cognitive functions and behavior, so it could be an interesting strategy to improve this disorder. The aim of the present study is to verify the effects of multiple components physical training and the consumption of omega 3 on behavior, cognitive functions and the serum levels of BDNF and IGF-1 in ADHD children. Thus, 68 ADHD children, between seven and fourteen years old will be selected. The volunteers will be randomly divided into four groups: Physical Training Group (PTG), Omega Group (OG), Omega and Physical Training Group (OPTG) and Control Group (CG). The protocol of the experiment will last three months in which the OPTG will make physical training and receive fish oil capsules, and the PTG will make only the physical training and receive a placebo of fish oil. The others groups will be oriented not to make any type of physical training, but the OG will receive fish oil capsule, and the CG will receive a placebo of fish oil. Behavioral and cognitive functions evaluations and blood analysis will be made at the beginning and at the end of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Children with ADHD: male, between seven and fourteen years old, sedentary, studing in a regular school.

Exclusion Criteria:

* Taking psychoactive medications, taking omega supplement.

Ages: 7 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos F Galduróz, Md PhD, Principal Investigator — Universidade Federal de São Paulo (UNIFESP)
Locations (1):
- Departamento de Psicobiologia, São Paulo, Brazil

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600

RESULTS

PARTICIPANT FLOW:
Groups:
- Omega-3: Take Omega-3 Only
- Sedentary (Control): The sedentary group will be oriented not to make any type of physical training for three months.
- Placebo + Physical Training: The omega 3 group will receive 2g per day of mineral oil during 90 days treatment
  Physical Training
- Omega 3 + Physical Training: The omega 3 group will receive 2g per day of fish oil during 90 days treatment
  Physical Training
Period: Overall Study
Arm/Group | Omega-3 | Sedentary (Control) | Placebo + Physical Training | Omega 3 + Physical Training
Started | 14 | 14 | 12 | 13
Completed | 11 | 13 | 12 | 11
Not Completed | 3 | 1 | 0 | 2
Not completed — Protocol Violation | 3 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Omega-3 Only: Omega 3: Capsules of omega 3, 1000mg / capsules. Administered 3 times a day.
- Sedentary (Control): The sedentary group will be oriented not to make any type of physical training for three months.
  Omega 3: Capsules of omega 3, 1000mg / capsules. Administered 3 times a day.
- Placebo + Phsycal Training: The omega 3 group will receive 2g per day of mineral oil during 90 days treatment
  Physical Training
- Omega 3 + Phsycal Training: The omega 3 group will receive 2g per day of fish oil during 90 days treatment
  Physical Training
- Total: Total of all reporting groups
Arm/Group | Omega-3 Only | Sedentary (Control) | Placebo + Phsycal Training | Omega 3 + Phsycal Training | Total
Number analyzed (Participants) | 14 | 14 | 12 | 13 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.27 (2.20) | 10.85 (2.03) | 10.36 (2.71) | 10.55 (2.94) | 10.5075 (2.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 00 | 00 | 00 | 00 | 0
  Male | 14 | 14 | 12 | 13 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 12 | 13 | 53
  Not Hispanic or Latino | 00 | 00 | 00 | 00 | 0
  Unknown or Not Reported | 00 | 00 | 00 | 00 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 14 | 14 | 12 | 13 | 53

OUTCOME MEASURES:

1. Primary Outcome: Conners Scale
Description: Scores on the Conners scale. Scores above 60 indicate ADHD. Minimum 0 and a maximum of 126.
Time Frame: 3 months
Population: Conners scale and the child stress scale (ESI)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omega-3 Only | Sedentary (Control) | Placebo + Phsycal Training | Omega 3 + Phsycal Training
Number analyzed (Participants) | 14 | 14 | 12 | 13
units on a scale | 36.64 (12.75) | 42.31 (12.10) | 40.08 (14.47) | 36.82 (7.91)
Statistical Analysis 1: Comparison: Omega-3 Only vs Sedentary (Control) vs Placebo + Phsycal Training vs Omega 3 + Phsycal Training; Test type: Other; p = 0.05, Chi-squared, Corrected; Mean Difference (Final Values) = 5

ADVERSE EVENTS:
Arm/Group | Omega-3 Only | Sedentary (Control) | Placebo + Phsycal Training | Omega 3 + Phsycal Training
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes